CLINICAL TRIAL: NCT01039506
Title: A Prospective Observational Study of the Efficacy and Safety of CPT-11 Based Regimens for UGT1A1 Genotype Guided Patients With Metastatic Colorectal Cancer
Brief Title: An Observational Study of CPT-11 Based Regimens and UGT1A1 Genotypes in Metastatic Colorectal Cancer (mCRC)
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Other Study IDs: TOP009-061; 090945 (Other: JAPIC ID)
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Metastatic Colorectal Cancer
Keywords: UGT1A1, irinotecan
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — white cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- UGT1A1 genotyped patients: UGT1A1 genotyped patients receive CPT-11 based regimens
  Interventions: Drug: CPT-11 based regimens

INTERVENTIONS:
Drug: CPT-11 based regimens
  Other Names: FOLFIRI, CPT-11+S-1, CPT-11

SUMMARY:
The purpose of this study is to examine the correlation between UGT1A1 genotypes and the efficacy of CPT-11 based regimens (FOLFIRI, CPT-11+S-1, CPT-11) for patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal cancer (adenocarcinoma)
* UGT1A1 genotyped patients
* Patients to receiving FOLFIRI, CPT-11+S-1 and CPT-11 alone therapy (with or without molecular targeted agents)

Exclusion Criteria:

* Contraindication of CPT-11
* Eastern Cooperative Oncology Group (ECOG) Performance Score (PS) 3-4
* Patients to receiving CPT-11 as adjuvant chemotherapy
* History of pelvic irradiation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer treated with CPT-11 based regimens (FOLFIRI, CPT-11+S-1, CPT-11) in clinical practice in Japan
Sampling Method: Probability Sample
Enrollment: 1376 (Actual)
Dates: Start 2009-10-15 (Actual); Primary Completion 2016-04-28 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Within 3 years
  Percentage of participants alive without disease progression

SECONDARY OUTCOMES:
Overall survival | At 3 years
  Percentage of participants alive at end of study
Time to treatment failure | Within 3 years
  Duration of time (in months) from treatment to failure
Response rate | from Day 1 (treatment) through disease progression (within 3 years)
  Percentage of participants with an objective response
Disease control rate | Within 3 years
  Percentage of participants with controlled disease
Safety events | Within 3 years
  Adverse events will be collected during treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Oncology, National Defense Medical College Hospital, Tokorozawa-shi, Saitama, Japan

IPD SHARING:
Plan to Share IPD: No